CLINICAL TRIAL: NCT04143035
Title: Hemodynamic Resuscitation and Monitoring in Early Sepsis
Acronym: HERMES
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tata Memorial Centre (Other)
Collaborators: Indian Society of Critical Care Medicine (Other)
Responsible Party: Principal Investigator, Sheila Nainan Myatra, Professor, Tata Memorial Centre
Other Study IDs: 3364
Record Dates: First submitted 2019-10-19; First posted 2019-10-29 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
"Hemodynamic Resuscitation and Monitoring in Early Sepsis (HERMES Study)" involves recording of patient's medical data related to that has been collected as part of his/her routine medical care in ICU.

Presently there is no data from Indian ICUs on the way patients in early sepsis are resuscitated and monitored. There may exist a wide variation in clinical practice. The investigators would like to conduct an observational study in various levels of Indian ICUs, to prospectively collect data on adult patients admitted to ICU with early sepsis in a 60-day window period. Investigator would like to study the hemodynamic resuscitation and monitoring performed in these patients. In addition, Investigator would like to identify factors associated with improved outcomes and achieving the goals of the sepsis bundles in one, three and six hours.

The objectives of the study is to capture the patient characteristics and hemodynamic resuscitation and monitoring practices in patients presenting with early sepsis and hypotension to Indian ICUs

Investigator plan to recruit 50 -100 centers nationwide. Each center will be asked to collect data from at least 10 patients in a maximum time window of 60 days. A convenience sample of minimum 500 patients presenting to ICU with suspected sepsis and hypotension will be taken.

Each Centre will guarantee the integrity of data collection and ensure timely completion of the case record forms. Each center will select a 60 day window period for patient recruitment. The start date may be anytime any time between 1st August to 15th October 2019. Therefore, the recruitment window period will end for a respective centre, anytime between 30th September and 14th December 2019, depending on the start date. All consecutive patients in the 60-day period will be screened and those eligible will be enrolled.

This is an ISCCM(Indian Society of Critical Care Medicine) Research Committee funded study. The ISCCM will fund the Principal Investigator for all expenses related software development, website hosting, secretarial assistance and miscellaneous expenses related to the conduct of the study, data analysis and publication. No funding will be given to the investigators from the various participating centers for contributing data.

DETAILED DESCRIPTION:
INTRODUCTION Septic shock is the most commonly occurring of all types of shock.The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) defines septic shock as a subset of sepsis in which particularly profound circulatory, cellular, and metabolic abnormalities are associated with a greater risk of mortality than with sepsis alone. Patients with septic shock can be clinically identified by a vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia. This combination is associated with hospital mortality rates greater than 40%.

The "sepsis bundle" has been central to the implementation of the Surviving Sepsis Campaign (SSC) from the first publication of its evidence-based guidelines in 2004 through subsequent editions. Developed separately from the guidelines publication by the SSC, the bundles have been the cornerstone of sepsis quality improvement since 2005. An updated version was published in 2016 "Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock". There is compelling nature of the evidence in the literature which demonstrates an association between compliance with bundles and improved survival in patients with sepsis and septic shock. This has led to the adoption of the SSC measures by the National Quality Forum (NQF) and other departments. The important relationship between the bundles and survival was confirmed in a publication from this initiative.

The Surviving Sepsis Campaign released an updated one-hour sepsis bundle, which combines recommendations listed in the three-hour and six-hour bundles. This includes 5 elements: 1. measuring lactate levels 2. obtaining blood cultures before administering antibiotics 3. administering broad-spectrum antibiotics 4. fluid resuscitation for hypotension or lactate level ≥ 4 mmol/L and 5. use of vasopressors for hypotensive during or after fluid resuscitation to maintain MAP ≥ 65 mm Hg.

Presently there is no data from Indian ICUs on the way patients in early sepsis are resuscitated and monitored. There may exist a wide variation in clinical practice.The Investigator would like to conduct an observational study in various levels of Indian ICUs, to prospectively collect data on adult patients admitted to ICU with early sepsis in a 60-day window period. Investigator would like to study the hemodynamic resuscitation and monitoring performed in these patients. In addition, investigator would like to identify factors associated with improved outcomes and fulfilling the goals of the one hour SSC bundles within one, three and six hours in patients with sepsis and septic shock.

OBJECTIVES

1. To capture the patient characteristics and hemodynamic resuscitation and monitoring practices in patient presenting with early sepsis and hypotension to Indian ICUs
2. To determine various factors associated with improved survival in patients with septic shock
3. To determine factors associated with achieving the 1 hour, 3 hour and 6-hour resuscitation goals of the sepsis bundle in patients with septic shock

METHODS Study design- Prospective observational multi-center national cohort study.

Patient Recruitment

ISCCM members across India will be contacted to register their ICUs in the study, through emails sent from the ISCCM Research committee. Repeated emails will be sent over a two-month period. Hospitals with more than one ICU can enroll each of their ICUs separately. Each ICU will need to contribute a minimum of 10 adult patients with sepsis and hypotension in a 60 day window period.

Each center will designate a maximum of two local coordinators (PI and Co-PI) who will provide scientific and structural leadership in their centers. They will ensure that all local necessary ethical and regulatory approvals are obtained before the start of patient inclusion.

Local coordinators will guarantee the integrity of data collection and ensure timely completion of the case record forms. Each center will select a 60 day window period for patient recruitment. The start date may be anytime any time between 1st August to 15th October 2019. Therefore, the recruitment window period will end for a respective centre, anytime between 30th September and 14th December 2019, depending on the start date. All consecutive patients in the 60-day period will be screened and those eligible will be enrolled.

Data Collection

1. There will be no direct patient contact or intervention. Local coordinators will guarantee the integrity of data collection and ensure timely completion of CRFs (case record forms). Date related to the following will be collected prospectively from the charts:
2. Patient demographic data e.g. age, sex, comorbidities, likely source of sepsis
3. Total number of ICU patients, patients with sepsis and septic shock admitted to the ICU in the 60 days period
4. Patient clinical examination findings and severity of illness
5. Details of hemodynamic monitoring and other systemic monitoring and therapy performed in ICU e.g. fluid bolus, vasopressor agents, monitoring devices used, hemodynamic variables measured, mechanical ventilation, dialysis etc. in the first 3 days of ICU admission
6. Antibiotics administered and details of microbiology examinations
7. Adjunct therapies initiated for sepsis
8. ICU, hospital and 28-day mortality

Sample size The primary endpoint of study was to determine the incidence of ICU mortality in patients with septic shock admitted to Indian ICUs. The sample size calculation was done on the basis of INDICAPS I(Indian Intensive Care Case Mix and Practice Patterns Study-I) Study data (IJCCM April 2016). In this study the ICU mortality incidence was found to be 45% in patients with septic shock. Assuming the incidence rate found in this study, a sample size of 401 produces a two-sided 95% confidence interval with a width equal to 0.100 when the sample proportion is 0.450. Sample size calculation was done using PASS software. To account for attrition, Investigator will take a sample size of at least 450 patients. Investigator plan to recruit 50 -100 centers nationwide. Each center will be asked to collect data from at least 10 patients, hence investigator should be able to meet this target of >450 patients.

Statistical analysis The primary objective of the study is to determine the patient characteristics and hemodynamic resuscitation and monitoring practices in patient presenting with early sepsis and hypotension to Indian ICUs which will be analyzed using descriptive statistics. To determine various factors associated with improved survival in patients with septic shock investigator will use the Fisher's exact test or Pearson's χ2 test. Univariable and Multivariable logistic regression models will be developed to assess the independent effects on ICU mortality. To determine factors associated with achieving the 1 hour SSC Sepsis resuscitation bundle in 1 hour, 3 hours and 6-hours in patients with sepsis and septic shock will be assessed by Fisher's exact test or Pearson's χ2 test. Univariable and Multivariable logistic regression models will be developed to assess the independent effects on ICU mortality of the 1 hour, 3 hour and 6-hour resuscitation goals of the sepsis bundle in patients with sepsis and septic shock. The overall performance of the internally validated model will be assessed using Nagelkerke's R2 (R squared in logistic regression). The higher Nagelkerke's R2, the greater the strength of the model. The ability of the models to identify ICU mortality will be quantified as the area under the receiver operating characteristic curve (AUC). The AUC ranges from 50% to 100%, indicating no discriminative capacity to perfect discriminative capacity. The agreement between predicted probabilities and observed frequencies of the outcome will be assessed by visually inspecting the calibration plot. Last, the Hosmer and Lemeshow goodness-of-fit statistic will be computed as a quantitative measure of accuracy. A high outcome of this statistic is related to a low p-value, which indicates a poor fit. All analysis will two sided, and significance will set at a p-value of 0.05. Statistical analyses will be performed using SPSS (the statistical package for social sciences) IBM Corp. Released 2017. IBM SPSS Statistics for Windows, Version 25.0. Armonk, New York: IBM Corp and R studio (version 1.2).

INSTITUTIONAL ETHICS COMMITTEE (IEC) APPROVAL The local hospital investigators should ensure that all necessary local ethical and regulatory approvals are obtained if required, before the start of the study in their institution.

CONSENT FOR DATA COLLECTION This is an observational study and involves capture of data from the patient charts. There is no direct patient contact or intervention, hence written, informed consent is not mandatory. However, if required by the institution, consent may be taken from the patients legally accepted representative (LAR). Sample short consent forms for patient data capture will be provided by the PI in English, Hindi and Marathi. This may be translated in various regional languages as required by the local investigator

STUDY FUNDING This is an ISCCM Research Committee funded study. The ISCCM will fund the Principal Investigator institution for all expenses related software development, website hosting, secretarial assistance and miscellaneous expenses related to the conduct of the study, data analysis and publication (against actual bills). No funding will be given to the investigators from the various participating centres for contributing data.

DATA STORAGE AND OWNERSHIP The Principal Investigator will have ownership of the data. The data will be stored in the Principal Investigators department at Tata Memorial Hospital, Mumbai for 10 years.

PUBLICATION AND AUTHORSHIP POLICY The main results of study will be published in a peer-reviewed medical journal. Authorship policy will follow the International Committee of Medical Journal Editors (ICMJE) recommendations. Authorship will be considered based on contributions the study design and protocol development, recruitment of patients, data acquisition and cleaning, analysis and interpretation of the data, manuscript writing and final approval of the version to be published and agreement to be accountable for all aspects of the work, in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

Steering Committee - Members of the Steering Committee will include 7 members from the Principal Investigators center and 8 -10 experts from across the country. They will be involved and provide active guidance from inception till publication of the study.

Writing committee and main author list - Members of the steering committee and Principal Investigator from the top 3 centers with highest number of patient recruitment.

The Principal Investigator and Co-Principal Investigator from each participating ICU will be in the list of study collaborators and their names will be in the publication. The names of all the investigators will be indexed in PubMed depending on the journal policy.

SECONDARY ANALYSES After publication of the primary results, on request, the pooled dataset will be available for investigators for secondary analysis, after judgment and approval of scientific quality and validity by the steering committee. Before submission, the final version of all manuscripts related to the study dataset must be approved by the steering committee. The members of the writing committee will be authors of the publications derived from the study dataset.

ELIGIBILITY:
Inclusion criteria

1. Adult patients (≥ 18 years old)
2. Presenting to ICU with suspected sepsis
3. Presence of hypotension (Systolic BP ≤ 90 mmHg / Mean arterial pressure (MAP) ≤ 65mmhg or patient with Systolic BP > 90 mmHg / MAP >65mmHg on vasopressor.

Exclusion Criteria

1. Patient likely to be in shock due to reason other than sepsis (e.g. cardiogenic or hemorrhagic shock)
2. Decision taken for not intubating / ventilating /aggressive resuscitation prior to ICU admission
3. Patient transferred from another ICU OR another hospital (only if stay >7 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to ICU with suspected sepsis and hypotension
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
ICU Mortality | throughout ICU stay till discharge (up to 2 months)
  Overall ICU Mortality due to septic shock with hypotension
Completing the elements of the one hour SSC sepsis bundle in one 1 hour | 1 hour after admission upto 60 days from the study start date in respective study site (60 days)
  Identify factors associated with improved outcomes and fulfilling the goals of the one hour Surviving Sepsis Campaign (SSC) bundles within one, three and six hours in patients with sepsis and septic shock and to identify compliance with the one hour SSC bundle guidelines The Surviving Sepsis Campaign released an updated one-hour sepsis bundle, which combines recommendations listed in the three-hour and six-hour bundles. This includes 5 elements: 1. measuring lactate levels 2. obtaining blood cultures before administering antibiotics 3. administering broad-spectrum antibiotics 4. fluid resuscitation for hypotension or lactate level ≥ 4 mmol/L and 5. use of vasopressors for hypotensive during or after fluid resuscitation to maintain MAP ≥ 65 mm Hg

SECONDARY OUTCOMES:
Hospital mortality | throughout the hospital stay till discharge in the respective study site (up to 3 months)
  Over all mortality during the hospital stay
28-day mortality | From ICU admission to 28 days in the respective study site (up to 3 months)
  Over all mortality from ICU admission day to till 28 day
Completing the elements of the one hour SSC sepsis bundle in one, three and six hours | 1 hour, 3 hour and six hour after admission upto 60 days from the study start date in the respective study site (60 days )
  Identify factors associated with improved outcomes and fulfilling the goals of the one hour Surviving Sepsis Campaign (SSC) bundles within one, three and six hours in patients with sepsis and septic shock and to identify compliance with the one hour, three hour and six hour SSC bundle guidelines The Surviving Sepsis Campaign released an updated one-hour sepsis bundle, which combines recommendations listed in the three-hour and six-hour bundles. This includes 5 elements: 1. measuring lactate levels 2. obtaining blood cultures before administering antibiotics 3. administering broad-spectrum antibiotics 4. fluid resuscitation for hypotension or lactate level ≥ 4 mmol/L and 5. use of vasopressors for hypotensive during or after fluid resuscitation to maintain MAP ≥ 65 mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Sheila N Myatra, MD, Principal Investigator — Tata Memorial Hospital, Parel, Mumbai-12
Locations (247):
- India (247):
  - AIIMS Patna, Patna, Bihar
  - All india institute of medical sciences, Patna, Bihar
  - Anant Institute of Medical Sciences, Jabalpur, Madhya Pradesh
  - Breach Candy Hospital Trust, Mumbai, Maharashtra
  - Criticare Hospital and Research Institute, Nagpur, Maharashtra
  - Galaxy care hospital, Pune, Maharashtra
  - Sanjeevan Hospital, Pune, Maharashtra
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - Eternal Hospital, Jaipur, Rajasthan
  - Kamlesh Kanwar Shekhawat, Udaipur, Rajasthan
  - Pims, Udaipur, Rajasthan
  - Sarvodaya hospital and research centre, Farīdābād, Uttar Pradesh
  - Fortune Hospital, Kanpur, Uttar Pradesh
  - Sir Sundar lal Hospital, IMS, BHU, Varanasi, Varanasi, Uttar Pradesh
  - Sir Sunderlal Hospital, Varanasi, Uttar Pradesh
  - Nayati Hospital - Trauma & Acute Care Centre, Agra
  - Purushottam das Savitri Devi Cancer center, Agra
  - Pushpanjali Hospital, Agra
  - Rainbow Hospitals, Agra
  - Saideep Healthcare and Research Pvt Ltd, Ahilyanagar
  - Narayana Multispeciality Hospital, Ahmedabad
  - Sterling hospital, Ahmedabad
  - Zydus Hospitals Ahmedabad, Ahmedabad
  - J N Medical College & Hospital, Aligarh
  - Ohm Trauma centre and critical care, Aligarh
  - Emc hospital, Amritsar
  - Fortis Escorts Hospital Amritsar, Amritsar
  - Kamalnayan Bajaj hospital, Aurangabad
  - Mgm Medical College Hospital and Medical Centre Research Institute(McRi), Aurangabad
  - Oriion Citicare Superspeciality Hospital, Aurangabad
  - Shraddha hospital and critical care center, Aurangabad
  - Bhagwan Mahaveer Jain Hospital, Bangalore
  - Columbiaasia Referral Hospital, Yeshwantpur, Bangalore
  - Cytecare Cancer Hospital, Bangalore
  - Health care Global (HCG), Bangalore
  - Shifaa hospital, Bangalore
  - Shri Ram Murti Smarak Institute of Medical Sciences, Bareilly
  - Geeta Hospital and research centre, Barnagar
  - Aster R V Hospital, Bengaluru
  - Manipal hospital, Bengaluru
  - Mazumdar Shaw Medical Center, Bengaluru
  - Regal Hospital, Bengaluru
  - St John's Medical College Hospital, Bengaluru
  - Vydehi Institute of Medical Sciences and Research Centre, Bengaluru
  - Apollo Hospitals, Bhubaneshwar
  - Amri hospital ICU -1, Bhubaneswar
  - AMRI Hospitals, Bhubaneswar
  - Amri Hospital, Bhubaneswar
  - Apollo Hospitals, Bhubaneswar
  - Apollo Hospital, Bhubaneswar
  - BR Life Kalinga Hispital, Bhubaneswar
  - Care Hospitals, Bhubaneswar
  - Care Hospital, Bhubaneswar
  - Gudage Hospital, Bidar
  - Apollo Hospital Icu-1, Bilāspur
  - Apollo Hospital, Bilāspur
  - Ayush Hospital, Bījāpur
  - K.M.Memorial hospital and research centre, Bokāro
  - PGIMER, Chandigarh
  - Apollo Hospitals Enterprise limited, Chennai
  - Billroth hospital, Chennai
  - Dr.Rela Institute and Medical Centre, Chennai
  - Mgm Healthcare Ltd., Chennai
  - Sri Ramachandra Hospital, Chennai
  - Sri Ramchandra Medical Centre, Chennai
  - Kovai Medical Center Hospital and Research, Coimbatore
  - Royal Care Super Speciality Hospital, Coimbatore
  - Ashwini Hospital, Cuttack
  - Goodluck Hospital, Cuttack
  - Scb Medical College and Hospital, Cuttack
  - SCB Medical College, Cuttack
  - Paras Global Hospital, Darbhanga
  - Dharmshila Narayana Superspeciality Hospital, Delhi
  - Dr. Ram Manohar Lohia Hospital ,New Delhi, Delhi
  - Dr. Ram Manohar Lohia Hospital, Delhi
  - kailash Hospital and heart Institute, Delhi
  - Pushpawati Singhania Research Institute, Delhi
  - Sir Ganga Ram Hospital, Delhi
  - BKL Walawalkar Hospital, Dervān
  - Muthukrishnan Periasamy, Erode
  - Qrg Healthcity, Faridabad
  - Yashoda super specialty hospital, kaushambi, Ghaziabad
  - City Hospital, Gorakhpur
  - Dr.Ramesh Cardiac and Multiplicity PVT LTD, Guntur
  - GBR super speciality hospitals, Guntur
  - Lalitha Super Specialities Hospital, Guntur
  - Samistha Hospital and Research Institute, Guntur
  - Apollo Hospitals Guwahati, Guwahati
  - Apollo hospitals, Guwahati
  - Ayursundra Superspecialty hospital, Guwahati
  - Dispur Hospitals pvt Ltd, Guwahati
  - Gnrc Hospitas, Dispur, Guwahati
  - Health City, Guwahati
  - Nemcare Hospital, Guwahati
  - Medanta Medicity, Gūrgaon
  - Medanta the medicity hospital, Gūrgaon
  - Medanta the medicity, Gūrgaon
  - Narayana Super Specialty Hospital, Gūrgaon
  - VPS Medeor Hospital, Gūrgaon
  - Santhi Hospital, Hosūr
  - Aig Hospitals, Gachibowli, Hyderabad
  - Apollo Health City ICU-1, Hyderabad
  - Apollo health city, Hyderabad
  - Aware Gleneagles Global Hospital, Hyderabad
  - Care hospital and institute of medical sciences, Hyderabad
  - Care hospitals banjara, Hyderabad
  - CENTURY hospital, Hyderabad
  - Century Super Speciality Hospital, Hyderabad
  - Continental Hospitals, Hyderabad
  - Gleneagles Global Hospital, Hyderabad
  - Krishna Institute of Medical Sciences, Hyderabad
  - Rainbow childrnes hospital, Hyderabad
  - South Central Railway Hospital ICU-1, Hyderabad
  - South Central Railway Hospital, Hyderabad
  - Virinchi Hospital, Hyderabad
  - Yashoda Hospital, Hyderabad
  - Choithram hospital, Indore
  - Dodeja Hospital, Jabalpur
  - Apex Hospital, Jaipur
  - Manipal hospital, Jaipur
  - Shubh Hospital, Jaipur
  - shrimann superspeciality hospital ICU-1, Jalandhar
  - Shrimann Superspeciality Hospital, Jalandhar
  - Kripa Critical Care and Trauma Centre, Jalgaon
  - Smvd Narayana Superspeciality Hospital, Jammu
  - Tata Main Hospital, Jamshedpur
  - All India Institute of Medical Sciences, jodhpur, Jodhpur
  - Ved Hospital, Kalyān
  - Abha superspeciality hospital, Kanpur
  - Regency hospital ltd tower 1, Kanpur
  - Shree krishna hospital ICU-1, Karamsad
  - Shree Krishna Hospital, Karamsad
  - Sankalpa hospital, Khammam
  - Amrita institute of Medical Sciences, Kochi
  - MOSC Medical College, Kochi
  - AMRI Hospital Mukundapur, Kolkata
  - AMRI Hospital, DHAKURIA, Kolkata
  - Apollo Gleneagles Hospital, Kolkata
  - Bellevue Clinic, Kolkata
  - Fortis Hospital Anandapur, Kolkata
  - Institute of Neurosciences Kolkata, Kolkata
  - Medica Superspecialty Hospital, Kolkata
  - Peerless Hospitex Hospital and Research Center Limited, Kolkata
  - Tata Medical Center, Kolkata
  - Travancore medical college,medicity, Kollam
  - Govt.Medical college, Kottayam
  - King George's Medical University, Lucknow
  - Christian Medical College, Ludhiana
  - Apollo speciality hospital, Madurai
  - Kasturba medical college, Manipal, Manipal
  - Nayati medicity hospital, Mathura
  - Manglam Hosp, Meerut
  - Metro Hospital and heart Institute, Meerut
  - Cheema Medical Complex, Mohali
  - Fortis Hospital, Mohali
  - MAX Superspecialty Hospital, Mohali
  - Asian Cancer Institute, Mumbai
  - Bhatia Hospital, Mumbai
  - Dr L H HIRANANDANI HOSPITAL, Mumbai
  - Fortis hiranandani hospital, Mumbai
  - Fortis Hospital Mulund, Mumbai
  - Fortis hospitals, Mumbai
  - Global Hospital,Parel, Mumbai
  - Global Hospital, Mumbai
  - Holy Family Hospital, Mumbai
  - Nanavati Hospital Icu-1, Mumbai
  - Nanavati hospital ICU-2, Mumbai
  - Nanavati Hospital Icu-3, Mumbai
  - Nanavati Hospital, Mumbai
  - Nanavati hosptial, Mumbai
  - Pd Hinduja National Hospital and Mrc, Mumbai
  - s.l.Rahej hospital- a fortis associate, Mumbai
  - Sir H N Reliance Foundation Hospital, Mumbai
  - Suasth Health Care, Mumbai
  - Tata Memorial Hospital (FICU), Mumbai
  - Tata Memorial Hospital (SICU), Mumbai
  - Wockhardt Hopsital South Mumbai, Mumbai
  - Cauvery Heart and multispeciality hospital, Mysore
  - Jss Hospital, Mysore
  - Gopalagowda Shanthaveri Memorial Hospital, Mysuru
  - Aditya Hospital, Nagpur
  - Dew medicare and Trinity Hospital, Nagpur
  - Dr V E Tambe Critical Care, Nagpur
  - Meditrina Institute Of Medical Scineces, Nagpur
  - Orange City Hospital And Research Institute, Nagpur
  - Rahate Surgical Hospital and Iccu, Nagpur
  - Shree Hospital and Critical Care Centre, Nagpur
  - Apollo Hospitals, Nashik
  - National Burns Centre, Navi Mumbai
  - Narayana Medical College Icu-1, Nellore
  - Narayana Medical College, Nellore
  - Simhapuri Hospital, Nellore
  - Batra Hospital & Medical Research Center, New Delhi
  - Batra Hospital, New Delhi
  - BLK hospital, New Delhi
  - Blk Superspeciality Hospital, New Delhi
  - Fortis Escorts Heart Institute, New Delhi
  - Fortis Hospital, Shalimar Bagh, New Delhi
  - GB Pant Institute of Post Graduate Medical Education & Research, New Delhi
  - Indraprastha Apollo Hospitals ICU-1, New Delhi
  - Indraprastha apollo hospitals, New Delhi
  - Max Super Specialty Hospital Patparganj, New Delhi
  - Northern railway central hospital, New Delhi
  - Sri balaji action medical institute ICU-1, New Delhi
  - Sri Balaji Action Medical Institute, New Delhi
  - Venkateshwar Hospital, New Delhi
  - Fortis Hospital, Noida
  - Promhex Multispeciality Hospital, Noida
  - Ojas hospital, Panchkula
  - All India Institute of Medical Sciences Patna, Patna
  - Indira Gandhi Institute of Medical Sciences, Patna
  - Prabhat Kumar, Patna
  - Bharati Vidyapeeth Deemed university and Medical College Hospital, Pune
  - Columbia Asia hospital, Pune
  - Jupiter Hospital, Pune
  - Niramaya Hoapital, Pune
  - Ruby Hall Clinic Icu-1, Pune
  - Ruby Hall Clinic ICU-2, Pune
  - Vishwaraj Hospital & Research Centre, Pune
  - Vishwaraj Hospital& Research Center, Pune
  - Om Hospital, Raipur
  - Pt. J. N. M. Medical College, Raipur
  - Ramskrishna care hospital, Raipur
  - Shree Narayana Hospital, Raipur
  - Genesis Multispeciality Hospital, Rajkot
  - Shree Giriraj Multispeciality hospital, Rajkot
  - Shree Giriraj Multispecialty Hospital, Rajkot
  - Sterling Hospital, Rajkot (A Division of Sterling Addlife India Private Limited), Rajkot
  - Synergy superspeciality hospital, Rajkot
  - Bhagwan Mahavir Medica Superspecialty Hospital, Ranchi
  - Sagarshree Hospital, Sāgar
  - Abdul Waheed Mir, Srinagar
  - Sheri Kashmir Institute of Medical Sciences, Srinagar
  - Kiran Hospital, Surat
  - Shree Sardar Smarak Hospital, Surat
  - Trichy Srm Medical College Hospital & Research Centre, Tiruchirappalli
  - Believers Church Medical College and Hospital, Tiruvalla
  - Kerala Institute of Medical sciences, Trivandrum
  - Siddaganga hospital and research centre, Tūmulūru
  - Sterling Hospitals, Vadodara
  - Homi Bhaba Cancer Hospital & Pandit Madan Mohan Malviya Cancer Centre,Tata Memorial Centre,Varanasi, Varanasi
  - S S Hospital BHU VARANASI, Varanasi
  - Christian Medical College, Vellore
  - Nagarjuna hospital, Vijayawada
  - St Ann Hospital, Visakhapatnam
  - Samraksha super speciality, Warangal
  - Arnam Hospital, Wardha

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available

REFERENCES:
- [Background] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Background] Dellinger RP, Carlet JM, Masur H, Gerlach H, Calandra T, Cohen J, Gea-Banacloche J, Keh D, Marshall JC, Parker MM, Ramsay G, Zimmerman JL, Vincent JL, Levy MM; Surviving Sepsis Campaign Management Guidelines Committee. Surviving Sepsis Campaign guidelines for management of severe sepsis and septic shock. Crit Care Med. 2004 Mar;32(3):858-73. doi: 10.1097/01.ccm.0000117317.18092.e4. PMID 15090974
- [Background] Dellinger RP, Carlet JM, Masur H, Gerlach H, Calandra T, Cohen J, Gea-Banacloche J, Keh D, Marshall JC, Parker MM, Ramsay G, Zimmerman JL, Vincent JL, Levy MM. Surviving Sepsis Campaign guidelines for management of severe sepsis and septic shock. Intensive Care Med. 2004 Apr;30(4):536-55. doi: 10.1007/s00134-004-2210-z. Epub 2004 Mar 3. PMID 14997291
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Intensive Care Med. 2008 Jan;34(1):17-60. doi: 10.1007/s00134-007-0934-2. Epub 2007 Dec 4. PMID 18058085
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Levy MM, Dellinger RP, Townsend SR, Linde-Zwirble WT, Marshall JC, Bion J, Schorr C, Artigas A, Ramsay G, Beale R, Parker MM, Gerlach H, Reinhart K, Silva E, Harvey M, Regan S, Angus DC; Surviving Sepsis Campaign. The Surviving Sepsis Campaign: results of an international guideline-based performance improvement program targeting severe sepsis. Crit Care Med. 2010 Feb;38(2):367-74. doi: 10.1097/CCM.0b013e3181cb0cdc. PMID 20035219
- [Background] Levy MM, Rhodes A, Phillips GS, Townsend SR, Schorr CA, Beale R, Osborn T, Lemeshow S, Chiche JD, Artigas A, Dellinger RP. Surviving Sepsis Campaign: association between performance metrics and outcomes in a 7.5-year study. Crit Care Med. 2015 Jan;43(1):3-12. doi: 10.1097/CCM.0000000000000723. PMID 25275252
- [Background] Levy MM, Pronovost PJ, Dellinger RP, Townsend S, Resar RK, Clemmer TP, Ramsay G. Sepsis change bundles: converting guidelines into meaningful change in behavior and clinical outcome. Crit Care Med. 2004 Nov;32(11 Suppl):S595-7. doi: 10.1097/01.ccm.0000147016.53607.c4. No abstract available. PMID 15542969
- [Background] Damiani E, Donati A, Serafini G, Rinaldi L, Adrario E, Pelaia P, Busani S, Girardis M. Effect of performance improvement programs on compliance with sepsis bundles and mortality: a systematic review and meta-analysis of observational studies. PLoS One. 2015 May 6;10(5):e0125827. doi: 10.1371/journal.pone.0125827. eCollection 2015. PMID 25946168
- [Background] Rhodes A, Phillips G, Beale R, Cecconi M, Chiche JD, De Backer D, Divatia J, Du B, Evans L, Ferrer R, Girardis M, Koulenti D, Machado F, Simpson SQ, Tan CC, Wittebole X, Levy M. The Surviving Sepsis Campaign bundles and outcome: results from the International Multicentre Prevalence Study on Sepsis (the IMPreSS study). Intensive Care Med. 2015 Sep;41(9):1620-8. doi: 10.1007/s00134-015-3906-y. Epub 2015 Jun 25. PMID 26109396
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Seymour CW, Gesten F, Prescott HC, Friedrich ME, Iwashyna TJ, Phillips GS, Lemeshow S, Osborn T, Terry KM, Levy MM. Time to Treatment and Mortality during Mandated Emergency Care for Sepsis. N Engl J Med. 2017 Jun 8;376(23):2235-2244. doi: 10.1056/NEJMoa1703058. Epub 2017 May 21. PMID 28528569
- [Background] Liu VX, Morehouse JW, Marelich GP, Soule J, Russell T, Skeath M, Adams C, Escobar GJ, Whippy A. Multicenter Implementation of a Treatment Bundle for Patients with Sepsis and Intermediate Lactate Values. Am J Respir Crit Care Med. 2016 Jun 1;193(11):1264-70. doi: 10.1164/rccm.201507-1489OC. PMID 26695114
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04143035/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT04143035/ICF_001.pdf